CLINICAL TRIAL: NCT06677697
Title: Comparative Study of 0.5% Bupivacaine and 0.5% Ropivacaine in Per Operative Continuous Lumber Epidural Anaesthesia of Lower Limb Bypass Surgery
Brief Title: Comparative Study of Bupivacaine and Ropivacaine in Lumber Epidural Lower Limb Bypass Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: ibrahim cardiac hospital and research institute (Other)
Collaborators: Bangladesh Institute of Research and Rehabilitation in Diabetes, Endocrine and Metabolic Disorders (Other)
Responsible Party: Principal Investigator, Raju Ahmed, Associate Professor, ibrahim cardiac hospital and research institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ICHRI/res/GA/2020/02; ICHRI/res/GA/2020/02 (Other: ICHRI)
Record Dates: First submitted 2024-10-29; First posted 2024-11-07 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Lower Limb Injuries
Keywords: Ropivacaine, Bupivacaine,; Epidural Anaesthesia,; Lower limb Bypass surgeries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group A 30 participant received 0.5% Bupivacaine (No Intervention): Group A 30 participant received 0.5% Bupivacaine
- Group B 30 participant received 0.5% rupivacaine (Experimental): Group B 30 participant received 0.5% rupivacaine
  Interventions: Drug: Ropivacaine 0,5%

INTERVENTIONS:
Drug: Ropivacaine 0,5% — Group B 30 patients recive 0.5% ropivacine
  Arms: Group B 30 participant received 0.5% rupivacaine

SUMMARY:
Regional anaesthesia is an important part in clinical anaesthesiology now a day. Epidural block is a commonly used regional technique alternative for general anaesthesia in case of lower limb bypass surgery. Bupivacaine and Ropivacaine both are amide local anaesthetics. This study was to compare the efficacy of 0.5% Bupivacaine with 0.5% Ropivacaine in lumber epidural block for lower limb bypass surgery. The aim of the study was to compare the hemodynamic changes and adverse effects between the two groups and the onset of sensory and motor blockade in lower limb bypass surgery.

Material and method: Sixty(60) patients with American Society of Anaesthesiologists class II/III scheduled for elective lower limb bypass surgeries were randomly allocated into two groups .Group B received 0.5% Bupivacaine, and group R received 0.5% Ropivacaine for epidural anaesthesia at the level of L4 & L5. The onset of sensory and motor block and adverse events during the peroperative period were noted.

DETAILED DESCRIPTION:
Introduction:

Epidural anaesthesia has been found to be a well-known technique for lower limb bypass surgeries as it provides effective sensory and motor blockade in an awake patient for longer duration. Moreover, Epidural anaesthesia provides better control of pain and satisfactory analgesia in postoperative period without any respiratory complications. Bupivacaine & Ropivacaine both are amide local anaesthetics. Bupivacaine being more cardiotoxic there has been paradigm shift to ropivacaine which is less cardiotoxic and widely used in epidural and spinal anaesthesia to obtain intraoperative and postoperative pain relief with lesser side effects. It has been seen that ropivacaine blocks the sensory fibres more effectively as compared to the motor fibre. In addition; ropivacaine has been shown to have vasoconstrictor properties.

Our goal in this prospective, single blind, randomized study was to compare the anaesthetic characteristics of 0.5% Ropivacaine with that of 0.5% Bupivacaine when administered epidurally for lower limb bypass surgery.

Materials & Methods

This randomized single-blind study was conducted from 1st January '2021 to 31st December '2022 at the department of Anaesthesiology, Ibrahim Cardiac Hospital and Research Institute, Shahbagh, Dhaka, Bangladesh. After institutional ethical committee approval and informed written consent, a total number of 60 adult patients were randomly allocated into two groups (n=30) using a computerized random number table. Patients with ASA physical status II & III, aged between 30 and 60 years, scheduled for lower limb bypass surgeries were enrolled in this study.

Exclusion criteria included local infection at the site of puncture, patients having any neurological deficit in the lower limb, severe hepatic, respiratory, hematological disorders and known allergy to study drugs.

Group B received 0.5% Bupivacaine, and group R received 0.5% Ropivacaine for Epidural Anaesthesia.

Preoperative assessment included detailed history, physical examination, systemic examination, airway assessment and routine investigations, such as hemoglobin, total blood cell count, differential white blood cell count, platelet count, blood glucose, blood urea and serum creatinine. ECG and X-ray were also performed. Preoperative baseline vital parameters were recorded. Intravenous line was secured with an 18G canula, and infusion was started. Premedication was given with inj. Ondansetron 4 mg iv, inj. Ranitidine 50 mg iv. After skin infiltration with 1% Lidocaine, the epidural space was identified with loss of resistance method at the L4 & L5 interspace in the midline with a 16-gauge Tuohy needle. With the bevel of the needle directed cranially a catheter was inserted 3-5 cm through the needle, then a 2 ml of test dose of the study drug was given. The patient was then placed supine and a further 12 ml of the study drug was administered over a 3-5 min period. Continuous epidural anaesthesia was maintained by 3-5 ml/h through syringe pump. Sensory and motor block were assessed at 5, 10, 15, 20, 30 minutes after injection, then at 30 minutes interval. Motor block was assessed by Bromage scale, and sensory block was assessed by the blunt end of a 27-gauge needle based on a dermatome chart. Heart rate, blood pressure, SPO2 were recorded every 5 minutes interval per operatively but data were analysis at 5 min, 15 min, 25 min, 35 min, 45 min, 60 min, 90 min, 120 min, 150 min, 180 min, 240 min, 300 min and 360 min interval. The following side effects were observed: nausea, vomiting, respiratory depression, shivering, and episode of hypotension (20% decreases in MAP in relation to baseline values), bradycardia (HR <50 beats/min), and hypoxemia (SpO2 <90%). If systolic blood pressure is <20% from base line or MAP <60 mmHg, IV ephedrine 5 mg was given incrementally. If the HR is <50 beats/min, 0.6 mg atropine sulfate was administrated. Other parameters like duration of onset of sensory and motor block were assessed.

ELIGIBILITY:
Inclusion Criteria:

Sixty patients who underwent lower limb surgery -

Exclusion Criteria:

non operative patients

-

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
compare the efficacy of drug | 6 months
  compare the efficacy of 0.5% Bupivacaine with 0.5% Ropivacaine in lumber epidural block for lower limb bypass surgery.

CONTACTS AND LOCATIONS:
Overall Officials: raju ahmed, Principal Investigator — ibrahim cardiac resech
Locations (1):
- Ibrahim Cardiac Hospital and Research Institute, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: No